CLINICAL TRIAL: NCT04714970
Title: Repetitive Transcranial Magnetic Stimulation on Appetite and Cognitive Function in Schizophrenia
Brief Title: rTMS on Appetite and Cognitive Function in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central South University (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WU2021TMS
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; rTMS; Appetite; Cognitive Function
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: 60 participants are randomized, through the predetermined random number list, into intervention group or sham stimulation group in equal.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTBS stimulation (Experimental): The participants randomized into experimental group will receive iTBS stimulation of dlPFC 5 times a day, with 1h interval between two stimulations, and for 5 continuous days.
  Interventions: Device: iTBS
- Sham stimulation (Sham Comparator): The participants randomized intoSham group will receive Sham stimulation, as the coil vertical to the brain surface, 5 times a day, with 1h interval between two stimulations, and for 5 continuous days.
  Interventions: Device: Shame stimulation

INTERVENTIONS:
Device: iTBS — Intermittent theta burst stimulation (iTBS) on left dlPFC. 90% RMT, 50Hz within train and 5Hz train for 2 second and rest for 8 second. 600 train and 200 second in total.
  Arms: iTBS stimulation
Device: Shame stimulation — TMS coil vertical to the brain surface, with same protocol as iTBS
  Arms: Sham stimulation

SUMMARY:
The weight gain and metabolic dysfunction has been vital conditions for individuals with schizophrenia. rTMS is a promising novel intervention, which have strong potentials on moderating increased appetite and cognitive deficits in schizophrenia, as it has been proved for the treatment of depression.

Therefore, the investigators designed this randomized controlled clinical trial to evaluate the efficacy and safety of rTMS, using iTBS pattern, on prevention and treatment for elevated appetite and cognitive deficiency in individual with schizophrenia.

DETAILED DESCRIPTION:
The weight gain and metabolic dysfunction has been vital conditions for individuals with schizophrenia. The cognitive function deficit has also been a major symptom for schizophrenia. However, metabolic dysfunction could further impair the cognition. rTMS is a promising novel intervention, which have strong potentials on moderating increased appetite and cognitive deficits in schizophrenia, as it has been proved for the treatment of depression.

Therefore, the investigators designed this randomized controlled clinical trial to evaluate the efficacy and safety of rTMS, using iTBS pattern, on prevention of the elevated appetite and cognitive deficiency in individual with schizophrenia. The intervention will last for 5 continuous days and the follow-ups are scheduled at baseline, 6days and 36days. The primary outcomes include the change of MCCB score, TFEQ score and EEG data. Secondary outcomes include the change of serum metabolic indexes and anthropometry indexes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia in accordance with DSM-5
* Commorbid with significant weight gain after antipsychotics
* Informed Consent

Exclusion Criteria:

* Diagnosed with other mental disease in accordance with DSM-5
* Comorbid with other severe physiological disease
* Used antipsychotic, antidepressants, mood stabilizer, or other psychoactive substances before
* Drug or alcohol abuse
* Pregnant or lactating
* Contraindication to rTMS

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of Appetite | Change from Baseline to 6days and 36days
  Three-Factor Eating Questionnaire
Change of MCCB | Change from Baseline to 6days and 36days
  The MATRICS™ Consensus Cognitive Battery
Change of ERP | Change from Baseline to 6days and 36days
  Food picture ERP recorded by EEG

SECONDARY OUTCOMES:
Change of fasting glucose | Change from Baseline to 6days and 36days
  in mmol/l
Change of fasting insulin level | Change from Baseline to 6days and 36days
  in mmol/l
Change of Triglyceride | Change from Baseline to 6days and 36days
  in mmol/l
Change of Total Cholesterol | Change from Baseline to 6days and 36days
  in mmol/l
Change of LDL | Change from Baseline to 6days and 36days
  in mmol/l
Change of HDL | Change from Baseline to 6days and 36days
  in mmol/l
Change of BMI | Change from Baseline to 6days and 36days
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, Prof, Principal Investigator — Central South University Psychiatry Department
Locations (1):
- Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No